CLINICAL TRIAL: NCT06620965
Title: A Comparison of the Effectiveness of PNF and Mulligan Mobilization Techniques with Classic Physiotherapy Modalities in People with Neck Pain
Brief Title: A Comparison of the Effectiveness of PNF and Mulligan Mobilization Techniques with Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Faruk Daniisman, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNFvsMULLIGAN
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Neck Pain
Keywords: Neck pain; Rehabilitation
MeSH Terms: conditions — Neck Pain | interventions — Muscle Stretching Exercises; Methods

STUDY DESIGN:
Intervention Model Description: There are two groups: the Mulligan group, which applies Mulligan mobilization techniques, and the PNF group, which applies PNF techniques.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mulligan Mobilization Group (Active Comparator): Mulligan mobilization techniques will be applied
  Interventions: Procedure: Mulligan Mobilization Technique
- PNF group (Active Comparator): Proprioceptive Neuromuscular Facilitation techniques will be applied
  Interventions: Procedure: Proprioceptive Neuromuscular Facilitation (PNF) Technique

INTERVENTIONS:
Procedure: Mulligan Mobilization Technique — NAGs (Natural Apophyseal Glides) involve passive oscillatory movements of a spinal facet joint in an anterocranial direction, performed with the patient seated. SNAGs (Sustained Natural Apophyseal Glides) maintain facet glides during active movements, aiming to reach the joint's end range. In SNAGs, the patient actively participates, and overpressure is applied at the end of movements to enhance the range of motion. Techniques include increasing rotation, lateral flexion, flexion, and extension. These were applied by a certified physiotherapist three times a week for four weeks, aiming to improve joint mobility without causing pain.
  Arms: Mulligan Mobilization Group
Procedure: Proprioceptive Neuromuscular Facilitation (PNF) Technique — Proprioceptive Neuromuscular Facilitation (PNF) Technique: PNF consists of four movement patterns in two diagonals:
  Flexion-left rotation and extension-right rotation Flexion-right rotation and extension-left rotation 3 PNF techniques were applied.
  Combined Isotonic Contractions: This technique involves concentric, eccentric, and stabilizing contractions of a muscle group (agonist). The goal is to increase active range of motion (ROM), strength, and improve control and coordination.
  Dynamic Stabilization (Stabilizing Reversal): This involves applying resistance in various directions to prevent movement, aiming to enhance dynamic stability, strength, and agonist-antagonist coordination.
  Hold-Relax Technique: This relaxation method involves isometric contractions against maximum resistance without movement to increase passive ROM and reduce pain. These were applied by physiotherapist three times a week for four weeks, aiming to improve joint mobility without causing pain.
  Arms: PNF group

SUMMARY:
The aim of this study is to compare the effectiveness of PNF (Proprioceptive Neuromuscular Facilitation) and Mulligan Mobilization techniques with classical physiotherapy modalities in individuals with neck pain.

DETAILED DESCRIPTION:
Forty individuals with neck pain aged between 18-55 years will be randomly divided into two groups, PNF and Mulligan group. Classical physiotherapy modalities will be applied to all individuals 5 days a week. PNF group will receive PNF techniques three days a week and Mulligan group will receive Mulligan mobilization techniques three days a week. Participants will be treated for 4 weeks. The pain level of the patients whose demographic data were recorded; Visual Analog Scale (VAS), pressure pain threshold; algometer, range of motion (ROM); universal goniometer, functionality; Neck Disability Index, kinesiophobia; Tampa Kinesiophobia Scale, quality of life; SF-36 Quality of Life Scale, mood; Beck Depression Inventory, cervical muscle performance level; cervical performance tests will be measured before and after treatment.

Post-treatment pain intensity, kinesiophobia and depression level; the effectiveness of pressure pain threshold, ROM, functionality, quality of life and cervical muscle performance level will be compared within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Complaint of neck pain for at least 3 months
* Volunteer between the ages of 18-55
* Receiving a diagnosis of chronic neck pain by a physician

Exclusion Criteria:

* Having undergone a surgical procedure for the spine
* Exercise therapy and/or physical therapy within the last 1 year
* History of fracture in the cervical region
* Radiculopathy, myelopathy (motor and sensory loss), or neurological impairment
* Presence of Cardiac Pacemaker
* Positive vertebrobasilar artery test
* Having a blood clotting disorder
* Presence of cancer
* Being diagnosed with rheumatoid arthritis
* Those with systemic diseases targeting the cervical region
* Presence of active infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | From enrollment to the end of treatment at 4 weeks
  The intensity of pain was assessed separately during rest and activity using the Visual Analog Scale (VAS). The patient was informed that on a 10 cm ruler, a score of 0 indicated no pain and a score of 10 represented the most severe pain imaginable, and was asked to mark the point that represented their pain level. The marked point was then measured in centimeters on the ruler and recorded as the pain intensity data.
Pressure pain threshold test | From enrollment to the end of treatment at 4 weeks
  In the pressure pain threshold assessment, algometer capable of measuring up to 200 Newtons with a precision of 0.1 Newton was used. The pressure application surface of the algometer was blunt and non-sharp, with a diameter of 1 square centimeter. The individual was seated in a relaxed posture, facing away from the physiotherapist during the measurement. Prior to the assessment, the painful tender area was identified through palpation based on the patient's guidance. Before the application, the individual was informed, and the compression pressure was gradually increased perpendicularly to the surface. The patient was asked to indicate the moment when the pressure sensation transitioned to pain. Three measurements were taken at one-minute intervals, and the average of these measurements was recorded as the pressure pain threshold value.
Assessment of Joint Range of Motion (ROM) | From enrollment to the end of treatment at 4 weeks
  Active cervical range of motion for flexion, extension, right-left rotation, and right-left lateral flexion was assessed by the researcher using a Universal Goniometer. The goniometer was positioned at the pivot point of each movement, and the individual was instructed to move their neck to its full extent. During the assessment, patients were asked to keep their feet on the ground, sit with their hands resting on their thighs, and maintain a neutral pelvis. Movements were performed at a steady pace with shoulders and back stabilized, and a 5-10 second rest in a neutral position was required after each movement.
  For cervical flexion and extension, the physiotherapist stood beside the individual, aligning the pivot with the acromion and following the ear's midline projection. For lateral flexion, the physiotherapist stood behind the individual, aligning the pivot with the C7 spinous process and following the cervical vertebrae's spinal protrusions.
Assessment of Functional Level | From enrollment to the end of treatment at 4 weeks
  To assess patients' functional levels, the Turkish version of the Neck Disability Index (NDI) was used. This test evaluates disability in daily life due to neck pain. Each section is scored from 0 to 5, with 5 indicating complete disability and 0 indicating no disability, resulting in a total of 6 possible scores. Scores range from 0 to 50. The 10-section test assesses the impact of pain on pain level, personal care, lifting, reading, headaches, concentration, work, driving, sleep, and recreational activities. Scores are categorized as follows: 0-4 indicates no disability, 5-14 indicates mild disability, 15-24 indicates moderate disability, 25-34 indicates severe disability, and 35 or above indicates complete disability.
  The test-retest reliability of the Turkish version, as assessed by Telci and colleagues, has an Intraclass Correlation Coefficient (ICC) value of 0.979, indicating excellent reliability.
Assessment of Kinesiophobia | From enrollment to the end of treatment at 4 weeks
  To measure fear of movement and re-injury in patients, the Tampa Scale for Kinesiophobia, developed by Kori and colleagues, was used. The Turkish version, adapted by Tunca-Yılmaz and their team in 2011, has demonstrated excellent test-retest reliability with an Intraclass Correlation Coefficient (ICC) of 0.806 (95% confidence interval = 0.720-0.867). The test comprises 17 questions, with scores ranging from a minimum of 17 to a maximum of 68. Higher scores indicate a higher level of kinesiophobia in the individual.
Assessment of Quality of Life | From enrollment to the end of treatment at 4 weeks
  Patients' health-related quality of life was assessed using the Turkish version of the Short Form-36 (SF-36), validated and reliability-tested by Koçyiğit and colleagues. Reliability was evaluated using Cronbach's alpha coefficients, which ranged from 0.7324 to 0.7612, indicating acceptable internal consistency. Item-total score correlations, which measure the relationship between each item and the total score, ranged from 0.4712 to 0.8872. Validity was assessed by examining correlations with other measures, with correlation coefficients ranging from 0.44 to 0.65.
  The SF-36 consists of 36 items across 8 subscales: physical function, social function, general health, vitality, mental health, pain, and role limitations due to physical and emotional problems. Each subscale is scored from 0 to 100, with higher scores indicating better quality of life.
Emotional State Assessment | From enrollment to the end of treatment at 4 weeks
  Patients' emotional state was evaluated using the Turkish version of the Beck Depression Inventory. The Turkish validity and reliability study was conducted by Hisli in 1988. Reliability analysis, including item analysis (r: 0.80) and split-half techniques (r: 0.74), showed good correlation coefficients. For validity, the correlation coefficient with the Minnesota Multiphasic Personality Inventory scale was r: 0.50 (moderate).
  The questionnaire consists of 21 items, each with 4 response options. Patients were asked to select the option that best describes how they felt over the past week. Each item is scored from 0 to 3, with a maximum possible score of 63.
Assessment of Muscular Endurance | From enrollment to the end of treatment at 4 weeks
  Cervical Flexors: To evaluate cervical flexors, the patient was instructed to lie supine. The physiotherapist placed their hand under the patient's occiput. The patient's head was positioned in flexion, approximately 2.5 cm off the surface, and held straight. The patient was asked to maintain this position as long as possible, and the duration was recorded in seconds. The timing was stopped and recorded when the patient could no longer maintain the position or if the flexion was disrupted.
  Cervical Extensors: For evaluating cervical extensors, the patient was positioned face down, with their arms at their sides and head hanging off the edge of the bed. The physiotherapist supported and positioned the patient accordingly. Once the patient achieved the correct position, the test and stopwatch were started simultaneously. The test ended and the duration was recorded in seconds when the patient lost the position.

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Danışman, Ph.D, Principal Investigator — Kahramanmaraş Sütçü İmam Univerisity
Locations (1):
- Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No